CLINICAL TRIAL: NCT03014869
Title: Comparison of High Flow Nasal Cannula and Noninvasive Positive Ventilation(NPPV) in Moderate Chronic Obstructive Pulmonary Disease Exacerbation(AECOPD)
Brief Title: High Flow Nasal Cannula vs NPPV in Moderate Chronic Obstructive Pulmonary Disease Exacerbation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Qingyuan Zhan, head of Pulmonary and Critical care medicine ward 4, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1304304-2
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: COPD Exacerbation
Keywords: COPD Exacerbation; High Flow Oxygen; Noninvasive Positive Ventilation; moderate
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High flow nasal cannula (Experimental): High flow nasal cannula(OptiflowTM); Flow 25-60 L/min is set according to patients' comfort; FiO2 is adjusted to maintain peripheral capillary oxygen saturation(SpO2) 90-95%; temperature is set at 37 degree centigrade.
  Interventions: Device: High flow nasal cannula
- Noninvasive positive ventilation (No Intervention): Parameters are set according to NPPV protocols

INTERVENTIONS:
Device: High flow nasal cannula — High flow nasal cannula (HFNC) is a new emerging noninvasive respiratory support technology, which mainly includes high flow (15-60 L/min) device, heating humidification device and nasal cannula for high flow. A large number of physiological studies confirmed that HFNC has the following critical physiological effects: promoting airway humidification, improving tolerance of treatment, reducing the physiological dead space on the upper respiratory tract, producing a certain level of positive end expiratory pressure (2-7 cmH2O), decreasing the work of breathing and so on.
  Other Names: High flow oxygen
  Arms: High flow nasal cannula

SUMMARY:
For moderate AECOPD(pH<7.35), several guidelines have strongly recommended NPPV as standard therapy, which can reduce the rate of intubation and mortality. A few previous studies have shown that HFNC can efficiently improve alveoli ventilation and breathing pattern in some severe AECOPD patients. Therefore, we hypothesize that HFNC is not inferior to NPPV for preventing endotracheal intubation in moderate AECOPD patients. To assess this hypothesis, we performed a multicenter, randomized, noninferiority trial of HFNV vs NPPV in moderate AECOPD patients.

DETAILED DESCRIPTION:
Recently, many clinical studies have showed that HFNC can be successfully used in patients with hypoxemic respiratory failure to improve the comfort, to attenuate respiratory failure and to decrease the rate of tracheal intubation and mortality. Although theoretically HFNC is a potential and ideal treatment for AECOPD patients, the related clinical researches are very few. It still needs to further evaluate the safety and efficacy of HFNC in patients with AECOPD. For moderate AECOPD(pH<7.35), several guidelines have strongly recommended NPPV as standard therapy, which can reduce the rate of intubation and mortality. A few previous studies have shown that HFNC can efficiently improve alveoli ventilation and breathing pattern in some severe AECOPD patients. Therefore, we hypothesize that HFNC is not inferior to NPPV for preventing endotracheal intubation in moderate AECOPD patients. To assess this hypothesis, we performed a multicenter, randomized, noninferiority trial of HFNV vs NPPV in moderate AECOPD patients.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD; 7.35>pH≥7.25，PaCO2>50 mmHg

Exclusion Criteria:

* contraindications for NPPV, such as thick sputum, cough weakness, hemodynamic instability, etc.; need to be intubated immediately; refuse to engage in the study; severe organ dysfunction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
endotracheal intubation demand rate | 90days

SECONDARY OUTCOMES:
actual endotracheal intubation rate | 90days

CONTACTS AND LOCATIONS:
Overall Officials: Qingyuan Zhan, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No